CLINICAL TRIAL: NCT02576925
Title: Development and Validation of a Predictive Score for the Ischemic Etiology of a Transient Diplopia
Brief Title: A Predictive Score for the Ischemic Etiology of a Transient Diplopia (VASCO-DIP)
Acronym: VASCO-DIP
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: MOA_2015-7
Record Dates: First submitted 2015-10-13; First posted 2015-10-15 (Estimated); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Diplopia
MeSH Terms: conditions — Diplopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Eligible patients: Adults having had a transient diplopia during the last 8 days.
  Interventions: Other: Clinical, ophthalmological and neurological evaluation

INTERVENTIONS:
Other: Clinical, ophthalmological and neurological evaluation — Clinical : questionnaire about the symptoms and about the vascular risk factors Imagery :Cerebral MRI, MRI angiography of the supra-aortic trunks, ECG, Holter, transthoracic echocardiography, Biology : blood count, erythrocytes sedimentation rate, C reactive protein Ophthalomogy : visual field, optical coherence tomography, retinography

SUMMARY:
The transient diplopias (TD) is defined by a short diplopia. Their etiology may be ophthalmological, neurological non-ischemic or of ischemic origin.

The difficulty is to recognize an ischemic mechanism which imposes emergency cares.

A clinical score could help the clinician to recognize the etiology of the TD .

ELIGIBILITY:
Inclusion Criteria:

* Transient diplopia (i.e. less than 24 hours) during the last 8 days

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults having had a transient diplopia during the last 8 days and seen at the fondation ophtalmologique Adolphe de Rothschild
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2015-09-24 (Actual); Primary Completion 2025-09-23 (Estimated); Study Completion 2025-12-23 (Estimated)

PRIMARY OUTCOMES:
Etiology, ischemic or not, of the initial transient diplopia | 3 months
  Questionnaire about the symptoms and about the vascular risk factors, cerebral MRI, MRI angiography of the supra-aortic trunks, ECG, Holter, transthoracic echocardiography, blood count, erythrocytes sedimentation rate, C reactive protein, visual field, optical coherence tomography, retinography and a new evaluation after 3 months.

SECONDARY OUTCOMES:
Incidence of new transient diplopia ischemic attacks during the 3 months of follow-up | 3 months
  Questionnaire about the symptoms and about the vascular risk factors, cerebral MRI, MRI angiography of the supra-aortic trunks, ECG, Holter, transthoracic echocardiography, blood count, erythrocytes sedimentation rate, C reactive protein, visual field, optical coherence tomography, retinography and a new evaluation after 3 months.
Incidence of diplopia ischemic strokes during the 3 months of follow-up | 3 months
  Questionnaire about the symptoms and about the vascular risk factors, cerebral MRI, MRI angiography of the supra-aortic trunks, ECG, Holter, transthoracic echocardiography, blood count, erythrocytes sedimentation rate, C reactive protein, visual field, optical coherence tomography, retinography and a new evaluation after 3 months.
Incidence of transient ischemic attacks, visual or not visual, during the 3 months of follow-up | 3 months
  Questionnaire about the symptoms and about the vascular risk factors, cerebral MRI, MRI angiography of the supra-aortic trunks, ECG, Holter, transthoracic echocardiography, blood count, erythrocytes sedimentation rate, C reactive protein, visual field, optical coherence tomography, retinography and a new evaluation after 3 months.
Incidence of ischemic strokes, visual or not visual, during the 3 months of follow-up | 3 months
  Questionnaire about the symptoms and about the vascular risk factors, cerebral MRI, MRI angiography of the supra-aortic trunks, ECG, Holter, transthoracic echocardiography, blood count, erythrocytes sedimentation rate, C reactive protein, visual field, optical coherence tomography, retinography and a new evaluation after 3 months.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Bichat, Paris
  - Fondation Ophtalmologique Adolphe de Rothschild, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No